CLINICAL TRIAL: NCT07260630
Title: Comparison of the Acute Effects of Stretching, Myofascial Release, and Instrument-Assisted Soft Tissue Mobilization in Individuals With Hamstring Tightness: Randomized Double-Blind Study
Brief Title: Acute Effects of Different Soft Tissue Techniques on Hamstring Tightness
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, BEYZA YAZGAN DAĞLI, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BYDTUBITAK-2024/1
Record Dates: First submitted 2025-07-06; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hamstring Shortness
Keywords: mobilisation; IASTM; myofascial release; stretching; functional performance; strength; range of motion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stretching Group (Active Comparator): Participants receive manual static hamstring stretching for 5 minutes in repeated intervals.
  Interventions: Other: Stretching Group
- Myofascial Release Group (Active Comparator): Participants will perform self-myofascial release using a vibrating foam roller applied to the hamstring muscles.
  Interventions: Other: Self-Myofascial Release
- Instrument-Assisted Soft Tissue Mobilization (IASTM) Group (Active Comparator): The concave edge of an IASTM tool will be used to apply pressure along the posterior thigh.
  Interventions: Other: Instrument-Assisted Soft Tissue Mobilization
- Control Group (No Intervention): Participants in the control group will not receive any therapeutic intervention.

INTERVENTIONS:
Other: Stretching Group — Manual static stretching applied to the hamstring muscle in five 30-second sets, with 30-second rest intervals. Total application time is 5 minutes.
  Arms: Stretching Group
Other: Self-Myofascial Release — Vibrating foam roller (38 Hz) used for self-myofascial release applied to hamstring muscles. Three sets of 30 seconds, with 30 seconds rest between sets.
  Arms: Myofascial Release Group
Other: Instrument-Assisted Soft Tissue Mobilization — Application of IASTM using a concave-edged tool over the posterior thigh for 5 minutes to increase tissue mobility and flexibility.
  Arms: Instrument-Assisted Soft Tissue Mobilization (IASTM) Group

SUMMARY:
Flexibility is one of the key components of health-related physical fitness and is influenced by various factors such as age, gender, joint structure, and muscle anatomy. Hamstring tightness can contribute to multiple lower extremity injuries. While traditional methods like stretching and myofascial release are commonly used to improve flexibility, instrument-assisted soft tissue mobilization (IASTM) has recently gained popularity. However, no studies in the current literature have compared the acute effects of these three methods in individuals with hamstring tightness. This study aims to compare the acute effects of stretching, myofascial release, and IASTM in individuals diagnosed with hamstring tightness (defined as <65° of hip flexion in the straight leg raise test without neurological findings).

DETAILED DESCRIPTION:
Hamstring tightness is a common musculoskeletal problem that can contribute to lower extremity injuries and functional limitations. Flexibility, one of the fundamental components of physical fitness, can be influenced by multiple factors including age, sex, joint structure, and muscle properties. Among various therapeutic approaches, static stretching and myofascial release are conventionally used to improve hamstring flexibility. More recently, instrument-assisted soft tissue mobilization (IASTM) has gained popularity for its potential to increase range of motion and reduce muscle tension more rapidly than traditional methods.

The study aims to identify which intervention is most effective in increasing hamstring flexibility acutely and will provide evidence to guide clinical decision-making in sports rehabilitation and injury prevention. Additionally, this research intends to fill a gap in the literature, as no prior study has directly compared these three methods in individuals with hamstring tightness.

This study is designed as a prospective, randomized, controlled, double-blind trial to compare the acute and short-term effects of three different manual therapy interventions such as static stretching, self-myofascial release using a vibrating foam roller, and IASTM on individuals with clinically diagnosed hamstring tightness. A fourth group will serve as the control group and will receive no intervention.

A total of 36 healthy participants, aged 18 to 30 years, with hamstring tightness confirmed via the Straight Leg Raise (SLR) test (hip flexion <65° without neurological findings), will be randomly assigned into one of four groups. Each group will consist of 9 participants. Interventions will be applied for approximately 5 minutes. Assessments will be conducted at four time points: baseline (pre-intervention), immediately after intervention, 12 hours post-intervention, and 24 hours post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 30 years
* Presence of hamstring tightness (Straight Leg Raise angle < 65°)
* No diagnosed chronic diseases
* Voluntary participation and signed informed consent

Exclusion Criteria:

* History of lower extremity trauma or surgery
* Symptoms radiating to one or both legs due to hamstring, spinal, or sciatic nerve injury
* Ankle instability
* Neurological findings during the straight leg raise test
* Presence of hyperalgesia, hematoma, varicose veins, or skin infection in the lower limb

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Hamstring Flexibility | From enrollment to the end of treatment at 1 weeks
  Hamstring flexibility will be evaluated using the passive and active Straight Leg Raise (SLR) test. An angle <65° indicates tightness. Change in hip flexion range will be measured at each time point.
Change in Knee Extension Angle | From enrollment to the end of treatment at 1 weeks
  With the hip maintained at 90° flexion in a supine position, the passive and active knee extension angle will be measured using a goniometer. This test assesses the passive extensibility of the hamstring muscles.

SECONDARY OUTCOMES:
Change in Hamstring Muscle Strength | From enrollment to the end of treatment at 1 weeks
  Maximal isometric hamstring muscle strength will be measured using a handheld dynamometer.
Change in Quadriceps Muscle Strength | From enrollment to the end of treatment at 1 weeks
  Maximal isometric quadriceps strength will be assessed to evaluate potential reciprocal inhibition effects.
Functional Performance - Vertical Jump Test | From enrollment to the end of treatment at 1 weeks
  Vertical jump performance will be measured to assess functional changes in lower extremity power.
Functional Performance - Single-Leg Hop Test | From enrollment to the end of treatment at 1 weeks
  Single-leg horizontal hop distance will be recorded to evaluate functional lower limb performance.
Subjective Perception - Global Rating of Change Scale | From enrollment to the end of treatment at 1 weeks
  Participants will rate their perception of change in hamstring flexibility using a 15-point Global Rating of Change Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No